CLINICAL TRIAL: NCT02994706
Title: A Prospective Pilot Study of Home Monitoring in Adults With Cystic Fibrosis (HOMECF)
Brief Title: A Study of Home Monitoring in Adults With Cystic Fibrosis (HOMECF)
Acronym: HOME-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart of England NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012135RM
Record Dates: First submitted 2014-07-16; First posted 2016-12-16 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home monitoring (Experimental): Home monitoring will involve participants recording their symptoms twice weekly on a modified mobile phone and recording their lung function twice weekly using a digital spirometer. This data will be automatically transmitted to the CF team and we will contact patients on the mobile phone if symptoms and/or lung function decline below a set threshold, suggesting the onset of a pulmonary exacerbation. We will contact patients within 24 hours of symptoms and/or lung function falling below this set threshold.
  Interventions: Procedure: Home Monitoring
- Clinical Care (Active Comparator): Throughout the study period, participants will attend outpatient clinic visits as usual and treatment with antibiotics as clinically indicated.
  Interventions: Other: Clinical Care

INTERVENTIONS:
Procedure: Home Monitoring — Participants selected to receive home monitoring, in addition to routine CF care, will be given a digital lung function monitor (spirometer) and a modified mobile phone.
  Arms: Home monitoring
Other: Clinical Care — Participants selected for this arm will continue to receive routine clinical care.
  Arms: Clinical Care

SUMMARY:
Cystic fibrosis (CF) is the most common fatal inherited condition in Caucasians, causing recurrent chest infections and premature death due to lung failure. When patients develop chest infections their symptoms usually slowly worsen over the course of several days to weeks. Due to this gradual onset, patients often seek medical attention several days or weeks after symptoms start to worsen. The Investigators believe that if they were able to monitor patients more closely they could diagnose and treat chest infections earlier and consequently improve health outcomes.

The HOMECF study aims to investigate whether home monitoring is beneficial for adults with CF. 100 subjects will be randomly allocated, 50 to receive home monitoring and 50 to receive routine clinical care for 12 months. Subjects receiving home monitoring will measure their lung function and symptoms twice weekly and this data will be transmitted to the medical team by means of a modified mobile phone.

the Investigators hypothesize that home monitoring will allow them to diagnose chest infections at an earlier stage and reduce hospital inpatient days. They will also assess the subjects' experience of receiving home monitoring, the impact on body weight and lung function and and conduct a full health economic analysis to assess value for money. They will also ask subjects to collect a urine sample once weekly to allow us to measure urinary levels of inflammatory markers.

Subjects will be recruited at the West Midlands Adult CF Centre in Birmingham. The research team are well placed to carry out the study because it is a large regional adult CF centre with an excellent record of conducting clinical research.

DETAILED DESCRIPTION:
The principal question being answered by this research study is:

1. Does home monitoring reduce the total number of inpatient hospital days in adults with cystic fibrosis (CF) compared to routine clinical care?

The secondary objectives of this research study are to assess:

1. The effect of home monitoring on lung function in adults with cystic fibrosis (CF)
2. The effect of home monitoring on requirement for antibiotics in adults with CF
3. The effect of home monitoring on nutritional status in adults with CF
4. The effect of home monitoring on health related quality of life in adults with CF
5. Costeffectiveness analysis comparing the home monitoring period with the routine clinical care period
6. The patient experience of receiving home monitoring in adults with CF
7. Whether urine levels of inflammatory markers correlate with symptoms and lung function in adults with CF

The aim of this study is assess whether home monitoring is beneficial for adults with cystic fibrosis. Overall, 100 subjects will be recruited at the West Midlands Adult Centre and randomly allocated in a 1:1 ratio to receive home monitoring or routine clinical care for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of CF
* age over 18 years
* the requirement for 1 or more admission to hospital to receive intravenous antibiotics over the preceding 24 months
* clinically stable at the time of recruitment
* Patients who give informed consent.

Exclusion Criteria:

* patients who are currently participating in another clinical trial (excluding observational studies)
* pneumothorax or lung surgery within the previous 3 months, eye surgery (e.g. cataract operation) in the previous 4 weeks (since these factors prevent measurement of spirometry)
* Sputum infection with Burkholderia cenocepacia or Mycobacterium abscessus
* Current diagnosis of active allergic bronchopulmonary aspergillosis (ABPA)
* Previous lung transplantation procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of inpatient hospital days in the home monitoring group compared to the routine clinical care group | up to 12 months

SECONDARY OUTCOMES:
Change in FEV1 in the home monitoring group compared to the routine clinical care group | up to 12 months
Change in FVC in the home monitoring group compared to the routine | up to 12 months
Days on oral and intravenous antibiotics in the home monitoring group compared to the routine clinical care group | Up to 12 months
Change in body weight in the home monitoring group compared to the routine clinical care group | Up to 12 months
Change in BMI in the home monitoring group compared to the routine clinical care group | Up to 12 months
Change in CFQ-R scores in the home monitoring group compared to the routine clinical care group | Up to 12 months
  The Cystic Fibrosis Questionnaire Revised version (CFQ-R) is a multiple choice and likert questionnaire split into two sections: Demographics and Quality of Life. Answers of 'Always' or similar are deemed a higher value than 'Never' or similar. The total score is gathered by calculating the amount of 'positive' and 'negative' answers - 'positive' answers are those that are lower values (e.g. never) than those that are higher values (e.g. 'always)
Health economic analysis measured by EQ-5D-5L | Up to 12 months
  The Euro Quality of Life (EQ5D) is a multiple choice questionnaire split onto sections including Mobility, Self-Care, Usual activities, Pain/Discomfort, and Anxiety/Depression. For each of these sections, it asks if a person always have issues, some issues or no issues (e.g. Mobility - I have no problems / I have some problems / I am confined to bed). The total score is gathered by calculating the amount of 'positive' and 'negative' answers - 'positive' answers are those that are lower values (e.g. I have no issues) than those that are higher values (e.g. I am confined to bed). There is also a scale, ranging from 0 (worst imaginable health) to 100 (best imaginable health) with 99 intervals in between whereby the patient marks where they feel their current health lays.
Health economic analysis measured by ICECAP-A | Up to 12 months
  The ICEpop CAPability measure for Adults (ICECAP-A) is a multiple choice questionnaire split onto sections including 'Feeling Settled and Secure, Love, Friendship and Support, Being Independent, Achievement and progress, and Enjoyment and pleasure. For each of these sections, it asks whether a person has no problem, some problems, many problems or total problem with a certain area (e.g. Being Independent - I can achieve in all aspects of my life / I can achieve in many aspects of my life / I can achieve in some aspects of my life / I am unable to be at all independent). The total score is gathered by calculating the amount of 'positive' and 'negative' answers - 'positive' answers are those that are lower values (e.g. I can achieve in all aspects of my life) than those that are higher values (e.g. I am unable to be at all independent).
Costs associated with caring for each participant and the cost of conducting the study in the home monitoring group compared to the routine clinical care group | Up to 12 months
Patient experience assessed by a semi-structured qualitative interview in the home monitoring group compared to the routine clinical care group | Up to 12 months
Levels of relevant urine biomarkers in the home monitoring group associated with pulmonary exacerbations | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Nash, MD, Principal Investigator — Heart of England NHS Foundation Trust
Locations (1):
- Birmingham Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nash EF, Choyce J, Carrolan V, Justice E, Shaw KL, Sitch A, Mistry H, Whitehouse JL. A prospective randomised controlled mixed-methods pilot study of home monitoring in adults with cystic fibrosis. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666211070133. doi: 10.1177/17534666211070133. PMID 35274585
- [Derived] Choyce J, Shaw KL, Sitch AJ, Mistry H, Whitehouse JL, Nash EF. A prospective pilot study of home monitoring in adults with cystic fibrosis (HOME-CF): protocol for a randomised controlled trial. BMC Pulm Med. 2017 Jan 23;17(1):22. doi: 10.1186/s12890-017-0366-x. PMID 28114922